CLINICAL TRIAL: NCT06437002
Title: Exploring the Full Body Representation in Anorexia Nervosa and Bulimia Nervosa
Acronym: FULLBR_ANBN
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Turin, Italy (Other); Open University (Other); Heriot-Watt University (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: 49C403
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anorexia Nervosa/Bulimia
MeSH Terms: conditions — Anorexia Nervosa; Bulimia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- anorexia nervosa restrictive/ANr
  Interventions: Behavioral: Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body
- anorexia nervosa binge-purging/ANbp
  Interventions: Behavioral: Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body
- bulimia nervosa/bn
  Interventions: Behavioral: Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body
- Health control/Hc
  Interventions: Behavioral: Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body

INTERVENTIONS:
Behavioral: Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body — The MMC will be used as a measure of MI and it is adapted for use in hands, feet, and the whole body as well as for online experimentation. The task is comprised of two conditions, MI, and motor execution, in which respectively participants will be asked to imagine and execute a movement sequence with both hands and feet and the whole body.
  Hand movements: index and thumb opposition; thumb extension from the fist; middle finger crossed on the index finger; and extension of the index and the little fingers.
  Foot movements: foot internal rotation, foot external rotation, foot dorsiflexion, and foot plantarflexion.
  Whole-body movements: take a small bow, lift arms over the head and stand on the tips of the toes (stretch), extend hands forward and lower the backside (squats) and a small jump.
  The types of movements required to be executed by participants are simple and do not require much energy. Therefore, people affected by AN and BN should be able to perform them without problems.

SUMMARY:
The ability to mentally recall a motor act without any overt movement is called motor imagery (MI). The movement simulation that occurs on a cognitive level can be seen as a way in which we express the mental representation of the body in action. MI tasks can be used as a proxy for the exploration of the mental representations of the body. Interestingly, MI tasks differ in the degree of action monitoring required to resolve the task. More in detail, we can allocate MI tasks along a continuum that goes from more implicit MI tasks (less action monitoring required for the resolution of the task) to more explicit MI tasks (more action monitoring required for the resolution of the task).

Eating disorders such as anorexia nervosa (AN) and bulimia nervosa (BN) are both characterized by body image distortion and impairments (i.e. overestimation of the perceived body), however, on a different state of the physical body: on one hand we have a highly malnourished body, on the other hand, we might have a healthy-looking body or an overweight body. As above mentioned, MI tasks can be used as a proxy for the exploration of the mental representations of the body and people affected by AN and BN show impairment on their imagined body. This means that people affected by AN and BN might respond differently when assessed for their MI abilities.

We hypothesize that people affected by AN might show greater impairment in their motor imagery abilities because of the greater discrepancy between the physical body (malnourished) and the mental body representation in comparison to people affected by BN, who usually have a health weight, even an altered body representation. Nevertheless, we might expect the alteration of body representation not strictly linked to the physical body dimensions, in the case of no difference between AN and BN. This would be of relevance for the creation of rehabilitative programs.

DETAILED DESCRIPTION:
The ability to mentally recall a motor act without any overt movement is called motor imagery (MI). The movement simulation that occurs on a cognitive level can be seen as a way in which we express the mental representation of the body in action. MI tasks can be used as a proxy for the exploration of the mental representations of the body. Interestingly, MI tasks differ in the degree of action monitoring required to resolve the task. More in detail, we can allocate MI tasks along a continuum that goes from more implicit MI tasks (less action monitoring required for the resolution of the task) to more explicit MI tasks (more action monitoring required for the resolution of the task).

Eating disorders such as anorexia nervosa (AN) and bulimia nervosa (BN) are both characterized by body image distortion and impairments (i.e. overestimation of the perceived body, however, on a different state of the physical body: on one hand we have a highly malnourished body, on the other hand, we might have a healthy-looking body or an overweight body. As above mentioned, MI tasks can be used as a proxy for the exploration of the mental representations of the body and people affected by AN and BN show impairment on their imagined body. This means that people affected by AN and BN might respond differently when assessed for their MI abilities.

Recent studies explored MI, through more explicit and more implicit MI tasks in people affected by eating disorders, such as AN and BN. For example, when it comes to more implicit MI tasks, Campione et al observed that people affected by AN and BN do not show a temporal advantage when mentally rotating pictured hands based on their own hands compared to other hand stimuli, as opposed to controls. Authors point out how people affected by eating disorders show an alteration of the MI process highlighting an alteration of body schema. Authors grouped AN and BN patients in their analysis without considering the responses about the psychiatric condition. Recently, in a work by Scarpina et al, authors observed how people affected by AN present altered MI processes independently from the level of awareness required since alterations emerged in the more implicit (i.e. laterality judgment tasks) and more explicit (i.e. Mental Motor Chronometry (MMC) tasks) tasks. Such evidence points out an alteration of the imagery process in AN and confirms what was observed also by Campione et al for people suffering from AN. Both studies focused their attention on hands only. In the study of Urgesi et al, when using the own-body transformation task (requiring left-right judgments on a schematic human figure that may be facing toward (front-facing) or away from the observers (back-facing)), authors observed a partial impairment (t-score calculated as patients' reaction times on accuracy ratios) of people affected by BN in resolving such a more implicit MI task: people with BN were impaired in providing laterality judgments on the front-facing human figure, wherein participants had to perform a mental transformation of their own body to assume the perspective of the body stimulus. Interestingly, this study focused its attention on the full body mental representation, but for a more implicit type of task only. Purcell et al, again, grouped AN and BN participants and compared their performance to controls at a more implicit MI task, which involves several body parts (i.e. sensitive body parts: abdomen, buttocks, thigh; controls body parts: shin, forearm, head). Participants were asked to execute a movement or to imagine executing the same movement (i.e. sizing a body part) involving the body parts above-mentioned. People affected by AN and BN required significantly more time to imagine tracing sensitive body parts compared to control body parts than healthy controls (HCs). Despite Purcell et al consider their task as more implicit, in our opinion, in this experiment a more explicit process of MI was assessed. That is because "participants were asked to execute a movement or to imagine executing the same movement", this means that the degree of action monitoring, grounding the task resolution, highly increased because participants were made aware of using their MI skills to solve the task (i.e. participants are openly asked to execute and imagine movements). When it comes to the full body, Guardia et al observe that people affected by AN overestimate their body size when asked to judge whether or not a door aperture is wide enough for them to pass through (i.e. first-person perspective). This does not happen for a third person present in the room with them. This shows an overestimation of the mentally represented body in AN. Lastly, in the work of Meregalli et al, authors compared acute AN (not differentiated by the type, restrictive or binge purging) and control in a series of MI-based tasks: results evidence that patients with AN displayed greater difficulty than control in explicitly imagining movements, in mentally rotating human figures, and in adopting a different egocentric visuospatial perspective. No significant differences were observed in an MMC-based task and the mental rotation of 3D objects. Overall, these previous pieces of evidence may suggest altered MI processes in individuals affected by eating disorders, such as AN and BN. Interestingly, literature reports stronger results for people affected by AN and BN when the resolution of more implicit MI-based tasks is considered, while for more explicit ones (i.e. MMC tasks) results do not seem clear-cut.

In previous studies patients were often grouped within a more generic "eating disorder sample", rather than considered by the diagnosis, such as AN (restrictive vs binge purging) and BN, and no comparison between the three was made (AN restrictive vs AN binge purging vs BN). However, the psychopathology behind these disorders is very different. More in detail, AN is characterized by i) restriction of energy intake relative to requirements, leading to a significant low body weight in the context of the age, sex, developmental trajectory, and physical health (less than minimally normal/expected, ii) intense fear of gaining weight or becoming fat or persistent behavior that interferes with weight gain, and iii) disturbed by one's body weight or shape, self-worth influenced by body weight or shape, or persistent lack of recognition of seriousness of low body weight. Moreover, we can distinguish between the restricting type (i.e. During the last 3 months has not regularly engaged in binge-eating or purging) and the binge-purging type (i.e. During the last 3 months has regularly engaged in binge-eating or purging). Differently, when it comes to BN, the condition is characterized by i) recurrent episodes of binge eating, as characterized by both eating, within any 2-hour period, an amount of food that is definitively larger than what most individuals would eat in a similar period of time under similar circumstances, and a feeling that one cannot stop eating or control what or how much one is eating, ii) recurrent inappropriate compensatory behaviors in order to prevent weight gain such as self-induced vomiting; misuse of laxatives, diuretics, or other medications; fasting or excessive exercise, iii) the binge eating and inappropriate compensatory behaviors occur, on average, at least once a week for 3 months, iv) self-evaluation is unjustifiability influenced by body shape and weight, v) the disturbance does not occur exclusively during episodes of AN. Moreover, despite both AN and BN are characterized by body image distortion and impairments (i.e. overestimation of the perceived body), this occurs in response to a different state of the physical body (i.e. highly malnourished body vs healthy-looking body/overweight body). In regards to such clinical differences, studies evaluating MI processes, especially when different body parts are involved (e.g. hands and the whole body as for previous studies), should consider each condition per se, AN restrictive, AN binge-purging, and BN.

We hypothesize that people affected by AN might show greater impairment in their motor imagery abilities because of the greater discrepancy between the physical body (malnourished) and the mental body representation in comparison to people affected by BN, who usually have a health weight, even an altered body representation. Nevertheless, we might expect the alteration of body representation not strictly linked to the physical body dimensions, in the case of no difference between AN and BN. This would be of relevance for the creation of rehabilitative programs.

ELIGIBILITY:
People affected by AN

Inclusion Criteria:

* Female;
* age between 18 and 55 years old;
* diagnosis of AN (restrictive and binge-purging type*), as per DSM V criteria (APA, 2013);
* BMI ≤ 17,5 Kg/m2;
* right-handed (i.e. Edinburgh Handedness Inventory (EHI) (Veale, 2014)).

  * Restricting type: During the last 3 months, the individual has not engaged in recurrent episodes of binge eating or purging behaviour (i.e. self-induced vomiting or the misuse of laxatives, diuretics, or enemas). This subtype describes presentations in which weight loss is accomplished primarily through dieting, fasting, and/or excessive exercise.
  * Binge-eating/purging type: During the last 3 months, the individual has engaged in recurrent episodes of binge eating or purging behaviour (i.e. self-induced vomiting or the misuse of laxatives, diuretics, or enemas).

Exclusion criteria:

* presence of motor impairments, such as: motor disorders, broken limbs, inability to move, amputation of limbs, etc… because of the nature of the tasks - see the section Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body;
* presence of neurological deficits, motor disorders, or somatosensory perception disorders (e.g. peripheral neuropathy); previous head injury;
* schizophrenia spectrum disorders and other psychotic disorders on an acute phase;
* pregnancy;
* heavy use of medication because of acute symptoms.

People affected by BN

Inclusion Criteria:

* female;
* age between 18 and 55 years old;
* diagnosis of BN, as per DSM V criteria (APA, 2013);
* BMI ≤ 17,5 Kg/m2 or BMI ≥ 30 Kg/m2;
* right-handed (i.e. EHI (Veale, 2014)).

Exclusion criteria:

* presence of motor impairments, such as: motor disorders, broken limbs, inability to move, amputation of limbs, etc… because of the nature of the tasks - see the section Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body;
* presence of neurological deficits, motor disorders, or somatosensory perception disorders (e.g. peripheral neuropathy); previous head injury;
* schizophrenia spectrum disorders and other psychotic disorders on an acute phase;
* pregnancy;
* heavy use of medication because of acute symptoms.

HCs - enrolled voluntarily

Inclusion Criteria:

* female;
* age between 18 and 55 years old;
* right-handed (i.e. EHI (Veale, 2014)).

Exclusion criteria:

* history of eating disorders or obesity in the past 5 years and currently;
* BMI ≤ 17,5 Kg/m2 or BMI ≥ 30 Kg/m2;
* presence of motor impairments, such as: motor disorders, broken limbs, inability to move, amputation of limbs, etc… because of the nature of the tasks - see the section Mental Motor Chronometry (MMC) Task Hands and Feet and Whole Body;
* presence of neurological deficits, motor disorders, or somatosensory perception disorders (e.g. peripheral neuropathy); previous head injury;
* schizophrenia spectrum disorders and other psychotic disorders on an acute phase;
* pregnancy;
* heavy use of medication because of acute symptoms.

Comparability between the four groups (AN restrictive vs AN binge-purging vs BN vs HCs) in terms of age and education will be guaranteed.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Female subjects affected by AN (restrictive and binge-purging type) and BN who will be hospitalized at the U.O. dei Disturbi del Comportamento Alimentare, San Giuseppe Hospital, Piancavallo (VCO), Italy will be selected and will be considered eligible for participation in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mental Motor Chronometry (MMC) | Immediately after the intervention/procedure
  Participants will watch a video of each movement and then will be asked to practice the movements. This will be followed by the MI condition for each body district. During the MI trials, participants will be asked to imagine performing the sequence of movements for each hand and each foot, five times, as quickly and as accurately as possible with their eyes closed. The whole-body movement trials will be imagined five times, but the block of trials will be repeated twice to ensure each body district is imagined the same number of times (e.g. imagery for the left limb was repeated for the right limb). After the MI condition participants will complete the motor execution task for each body district.
  The order of the body district will be randomized between participants. For each participant and each body district, we will compute the average duration of the four movements for the right and the left side separately, both in the imagery and in the motor execution conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- istituto Auxologico italiano IRCSS, Milan, MI, Italy